CLINICAL TRIAL: NCT05164965
Title: C-reactive Protein and Homocysteine and Their Interaction Contribute to Postoperative Delirium
Brief Title: C-reactive Protein，Homocysteine，Postoperative Delirium
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Yuan Shen, MD, PhD, Chief of Psychiatry, Shanghai 10th People's Hospital
Other Study IDs: dsyy007
Record Dates: First submitted 2021-09-10; First posted 2021-12-21 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate how C-reactive protein (CRP) and homocysteine and their interaction contribute to postoperative delirium, based on our previous finding on the interactions of CRP, homocysteine and postoperative delirium.

DETAILED DESCRIPTION:
Postoperative delirium is a common complication of patients who undergo major surgery. It is frequently accompanied by adverse outcomes like Alzheimer's disease, high risk of postoperative complications and poor long-term outcomes, but its pathogenesis and biomarkers remain undetermined. Neuroinflammation is emerging as a popular hypothesis of developing postoperative delirium, particularly via microglial activation and increased pro-inflammatory cytokines in the brain. However, not every patient with surgery-induced inflammation develops postoperative delirium. Thus, inflammation alone may be insufficient to explain postoperative delirium. Patients who develop postoperative delirium may have other changes (predisposing factors) that exacerbate surgery-induced inflammation (precipitating factor), leading to neuronal dysfunction.

A potential predisposing factor is hyperhomocysteine, a pathogenesis implicated in cardiovascular and Alzheimer's disease. Previous studies had indicated that preoperative hyperhomocysteine may be related to postoperative delirium, but the findings are conflicting. More importantly, the interaction between inflammation and hyperhomocysteine remains unknown, which may contribute more to postoperative delirium than the inflammation alone or hyperhomocysteine alone.

Thus, this study is a prospective observational cohort study to evaluate the interaction between CRP and hyperhomocysteine and their contribution to postoperative delirium. Patients scheduled for orthopedic surgeries will be included. Written informed consent will be obtained from all the patients.

Preoperative assessments：Participants recruited will receive preoperative assessments one day before the scheduled surgery by two well-trained researchers. The assessments include demographic characteristics (e.g., age, sex, education, marital status )，age-adjusted Charlson comorbidity index (ACCI) , cognitive function assessments (mini-mental state examination [MMSE] and Confusion Assessment Method [CAM]). And similarly venous blood samples of patient will be collected for homocysteine and C-reactive protein measurements.

Outcome measurement： Postoperative delirium will be assessed for the first, second and third day after surgery (twice daily, in the morning and afternoon respectively) using the CAM and CAM-Severity (CAM-S) long-form by two trained assessors. And venous blood samples of patients will be collected after the anesthesia/surgery for C-reactive protein measurements.

ELIGIBILITY:
Inclusion Criteria:

1. were 60 years old or older
2. had a normal cognitive function at the time of enrollment, evidenced by a mini-mental state examination (MMSE) score above an education-adjusted threshold (18 for individuals with no school education, 20 for 1-6 years of education, or 24 for 7 or more years of education 27)
3. spoke Mandarin Chinese
4. were able to provide informed consent
5. scheduled for orthopaedic surgeries

Exclusion Criteria:

1. pre-existing delirium assessed according to the Confusion Assessment Method (CAM) algorithm;
2. prior neurologic diseases (Parkinson's disease, multiple sclerosis or stroke) according to the International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10);
3. history of mental disorders, e.g., major depressive disorder and schizophrenia, according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV);
4. unwillingness to comply with the assessments.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 60 years old or older and scheduled for orthopedic surgeries with an expected duration ≥ 2 h
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 3 days after surgery
  Incidence of postoperative delirium on postoperative day 1, 2 and 3 will be defined according to the confusion assessment methods (CAM).

SECONDARY OUTCOMES:
Severity of postoperative delirium | 3 days after surgery
  Severity of postoperative delirium on postoperative day 1, 2 and 3 will be defined according to he Confusion Assessment Method based delirium severity evaluation tool (CAM-S).The sum score of CAM-S ranges from 0 (no) to 19 (most severe).

OTHER OUTCOMES:
Pain Scores | 3 days after surgery
  Patient reported pain assessments would be performed using the Visual Analogue Scale (VAS), which ranging from 0 (without pain) to 10 (extremely painful) scores. Patients would be requested to report pain scores when they were resting and moving during 1-3 days after surgery, once daily. Both the worst score and average score over time would be reported.
Sleep difficulty | 3 days after surgery
  Patients self-reported sleep difficulty (including difficulty falling asleep, difficulty waking up and falling back asleep, waking up too early in the morning and sleepiness during the day) would be recorded for further analysis. Patients would be requested to report whether such sleep difficulty is newly emerging or re-emerging during 1-3 days after surgery, once daily. The rate of newly emerging sleep disorder would be report.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shen, MD, PhD, Principal Investigator — Shanghai, Shanghai, China, 200072
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No